CLINICAL TRIAL: NCT01198327
Title: Extended Follow-up of Patients With Macular Edema Due to bRanch rETinal Vein Occlusion (BRVO) or centrAl Retinal veIn occlusioN (CRVO) Previously Treated With Intravitreal Ranibizumab
Brief Title: Extended Follow-up of Patients With Macular Edema Due to Retinal Vein Occlusion
Acronym: RETAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peter A Campochiaro, MD (Other)
Collaborators: The Macula Foundation, Inc. (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Peter A Campochiaro, MD, Principal Investigator, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00040287
Record Dates: First submitted 2010-08-31; First posted 2010-09-10 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-11

CONDITIONS: Retinal Vein Occlusion
Keywords: RVO; CRVO; BRVO; Horizon; Bravo; Cruise
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab; zorubicin; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab as needed (Experimental): Intravitreal ranibizumab, .5mg dose, PRN but not less than 21 days apart; with optional peripheral laser to areas of non-perfusion.
  Interventions: Drug: ranibizumab; Other: Peripheral Laser

INTERVENTIONS:
Drug: ranibizumab — Intravitreal ranibizumab, .5mg dose, PRN but not less than 21 days apart.
  Other Names: RBZ, lucentis
Other: Peripheral Laser — Areas of nonperfusion identified on wide field angiograms will receive laser, if the patient is continuing to require ranibizumab injections.
  Other Names: Laser

SUMMARY:
This study evaluates long-term safety in patients with macular edema due to Retinal Vein Occlusion (RVO) originally enrolled in the BRAVO & CRUISE trials and subsequently followed in the HORIZON extension trial.

DETAILED DESCRIPTION:
There is strong evidence that ranibizumab provides benefit in subjects with macular edema due to RVO; however, some subjects required continued injections for years to maintain those benefits. It is likely that such subjects have continued production of VEGF (Vascular Endothelial Growth Factor) from areas of nonperfused retina in the periphery. One strategy is to perform scatter photocoagulation to areas of nonperfusion to reduce continued production of VEGF, but it is important to know if visual benefits are maintained when this is done, because if it is not, it would be better to continue intermittent injections of ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age greater than or equal to 18 years
* Completion of 12 months in BRAVO or CRUISE trials, with subsequent follow-up in the HORIZON extension study. Exit from HORIZON should be within 90 days of enrollment

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any condition that the investigator believes would pose a significant hazard to the subject if investigational therapy were initiated.
* Inability to comply with study or follow up procedures
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (6):
- United States (6):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Consultants Medical Group, Sacremento, California
  - Southeast Retina, Augusta, Georgia
  - Ophthalmic consultants of Boston, Boston, Massachusetts
  - Retina Associates of New Jersey, Teaneck, New Jersey
  - Retina Consultants of Houston, Houston, Texas

REFERENCES:
- [Background] Campochiaro PA, Hafiz G, Channa R, Shah SM, Nguyen QD, Ying H, Do DV, Zimmer-Galler I, Solomon SD, Sung JU, Syed B. Antagonism of vascular endothelial growth factor for macular edema caused by retinal vein occlusions: two-year outcomes. Ophthalmology. 2010 Dec;117(12):2387-2394.e1-5. doi: 10.1016/j.ophtha.2010.03.060. Epub 2010 Jul 13. PMID 20630595
- [Background] Campochiaro PA, Heier JS, Feiner L, Gray S, Saroj N, Rundle AC, Murahashi WY, Rubio RG; BRAVO Investigators. Ranibizumab for macular edema following branch retinal vein occlusion: six-month primary end point results of a phase III study. Ophthalmology. 2010 Jun;117(6):1102-1112.e1. doi: 10.1016/j.ophtha.2010.02.021. Epub 2010 Apr 15. PMID 20398941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 retinal vein occlusion patients from the HORIZON study(NCT01198327)were enrolled from 7 sites for long term follow up. The sites were: Wilmer Eye Institute, Ophthalmic Consultants of Boston, Retina Consultants of New Jersey, Retina Consultants Macula Group,Retina Consultants of Houston, Southeast Retina and Retina Vitreous Associates
Groups:
- Ranibizumab as Needed: Ranibizumab as needed, with optional peripheral laser to areas of non-perfusion.
Period: Overall Study
Arm/Group | Ranibizumab as Needed
Started | 66
Completed | 56
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab as Needed
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Serious Adverse Events.
Description: Record the serious adverse events, both ocular and non-ocular to gather long-term safety data.
Time Frame: 24 mos
Measure: Number; unit: number of serious adverse events
Arm/Group | Ranibizumab as Needed
Number analyzed (Participants) | 66
number of serious adverse events | 17

2. Secondary Outcome: Mean Changes in Visual Acuity
Description: Mean changes in visual acuity. Visual acuity is measured using standard ETDRS (Early Treatment Diabetic Retinopathy Study) charts which measure visual acuity in terms of letters( ETDRS Letters) read at a distance of 4 meters away from the chart. The ETDRS letters Score can be from 0 to 100, with 0 representing poor vision and 100 representing best vision.
Time Frame: 24 mos from study baseline
Measure: Mean (Standard Deviation); unit: ETDRS letters
Groups:
- Ranibizumab as Needed -CRVO: Ranibizumab as needed, with optional peripheral laser to areas of non-perfusion. CRVO stands for Central retinal vein occlusion.
- Ranibizumab as Needed -BRVO: Ranibizumab as needed, with optional peripheral laser to areas of non-perfusion. BRVO stands for branch retinal vein occlusion.
Arm/Group | Ranibizumab as Needed -CRVO | Ranibizumab as Needed -BRVO
Number analyzed (Participants) | 28 | 28
ETDRS letters | 14.0 (20.9) | 20.1 (17.2)

3. Secondary Outcome: Mean Change in Retinal Thickness
Description: Mean change in retinal thickness as measured by OCT (Optical Coherence Tomography).
Time Frame: 24 mos from study baseline
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Ranibizumab as Needed -CRVO | Ranibizumab as Needed -BRVO
Number analyzed (Participants) | 28 | 28
microns | -426.0 (270.1) | -236.2 (230.3)

ADVERSE EVENTS:
Arm/Group | Ranibizumab as Needed
Serious Adverse Events (participants affected / at risk) | 17/66
Other Adverse Events (participants affected / at risk) | 53/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab as Needed (N=66)
Death resulting from pre-existing idiopathic pulmonary fibrosis (General disorders) | 1 (1)
Death of unknown cause (General disorders) | 1 (1) — Reason for death could not be found out, despite multiple attempts to contact family members.
ECG for elective knee surgery showed inverted T waves, patient asymptomatic, admitted for workup (Cardiac disorders) | 1 (1) — Coronary artery bypass surgery, recovered
Mild chest discomfort for 6 mos, coronary angiography showed 2 obstructions (Cardiac disorders) | 1 (1) — Elective placement of 2 stents without complications, recovered
Tachycardia and went to the emergency department (Cardiac disorders) | 1 (1) — Cardioverter defibrillator implanted, recovered
Syncope with fall because of arrhythmia (Cardiac disorders) | 1 (1) — Pacemaker implanted, recovered
Chronic atrial fibrillation, CVA; bladder cancer identified during hospitalization (General disorders) | 1 (1) — Pacemaker implanted, administered anticoagulants,underwent surgery for bladder cancer; recovered
Head injury resulting from fall (General disorders) | 1 (1) — Received staples for scalp laceration, recovered
Urinary tract infection leading to septic shock (Infections and infestations) | 1 (1) — Hospitalized, recovered
Hospitalized for pneumonia (Infections and infestations) | 2 (3) — Recovered
Hospitalized for elective surgery (Musculoskeletal and connective tissue disorders) | 2 (3) — Recovered
Vitreous hemorrhage, (Eye disorders) | 1 (1) — resolved spontaneously
Second branch retinal vein occlusion in same eye (Eye disorders) | 1 (1) — Patient with an inferior branch retinal vein occlusion had resolution of edema, but a superior branch vein occlusion developed 27 months after last ranibizumab injection. Had severe ischemia, and neovascular glaucoma developed.
Retinal tear in a patient with branch retinal vein occlusion who did not receive any treatment (Eye disorders) | 1 (1)
Severe reaction to povidon-iodine (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab as Needed (N=66)
Upper Respiratory Infection (General disorders) | 20 (26) — This adverse event was specified as "Upper respiratory Infection". It was reported if a study subject had a common cold, viral bronchitis or sinusitis.
Ocular discomfort (Eye disorders) | 13 (15) — Discomfort after intravitreal injection
Subconjuctival Hemorrhage (Eye disorders) | 13 (21)
Vitreous Hemmorhage (Eye disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No